CLINICAL TRIAL: NCT05425342
Title: iECG: A Feasibility Study for Recording Chest Leads Using a Smartwatch Coupled With a Digital Image Processing Algorithm
Brief Title: iECG: Recording Chest Leads Using a Smartwatch With a Digital Image Processing Algorithm
Acronym: iECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2020-02470
Record Dates: First submitted 2020-12-08; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Electrocardiogram
Keywords: Electrocardiogram ECG; Smartwatch ECG; Wearables; eHealth; medical image processing; machine learning; self health check-up; telemedicine; digital medicine; bipolar chest leads; electrical signal quality; self-recordable smartwatch ECG; heart rhythm; cardiac pathology in ECG

STUDY DESIGN:
Intervention Model Description: single group, open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECG single group (Experimental): Patients will be instructed how to record an ECG on a smartwatch using the front camera of an iPad. In a second step, a standard ECG will be recorded by medical staff. The ECGs will then be compared by two board certified cardiologists
  Interventions: Device: Smartwatch ECG

INTERVENTIONS:
Device: Smartwatch ECG — Self-recorded 9-lead smartwatch ECGs

SUMMARY:
The purpose of this study is to evaluate the feasibility of a new method for self-recordable ECGs using a smartwatch coupled with an image processing algorithm. The long-term goal of this project is to establish such a method and to potentially integrate it into telemedical care.

DETAILED DESCRIPTION:
There is an increasing availability of smartwatches worldwide. Health-related features of these wearables such as heart rate and -rhythm analysis have become increasingly recognised. Some smartwatches are capable of recording an electrocardiogram (ECG) which yields important information about electrical heart activity. Recording a complete ECG with a smartwatch is challenging if the user has no prior medical experience. In this feasibility study we introduce a novel image processing tool that instructs the user to record an ECG using the front camera of an iPad. In a second step, a standard ECG will be recorded by medical staff. The ECGs will then be compared by two board certified cardiologists. The aim of the study is to evaluate the feasibility of self-recorded smartwatch ECGs. If this method can be established, it could markedly expand the diagnostic options for heart and vascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Participant ≥ 18 years
* Ability to record a smartwatch ECG
* Written informed consent as documented by signature from the participant

Exclusion Criteria:

* Smartwatch ECG or conventional ECG cannot be recorded due to comprehensible reasons (allergic reactions, wounds, etc.)
* Unable or not willing to sign informed consent
* Significant mental or cognitive impairment that could interfere with the measurements (e.g.

delirium, acute psychotic episode, etc., assessed by recruiting physician)

· Prior knowledge or experience in recording ECGs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Correctly recorded smartwatch ECG lead by patient | 1 hour
  The number of correctly recorded limb (I, II, III) and chest leads (bV1-bV6 where the letter "b" denotes bipolar chest leads) will be assessed. A correctly recorded lead is defined as a complete, 30-second long bipolar electrical signal obtained by the patient with the smartwatch afterpreviously being instructed. The number of correctly recorded smartwatch ECG leads is a measure to determine the feasibility of the method.

SECONDARY OUTCOMES:
Correctly identified chest lead position (V1-V6 vs. bV1-bV6) | 1 hour
  Chest ECG leads obtained with a traditional ECG (V1-V6) will be compared with the ones recorded with a smartwatch (bV1-bV6). The percentage of correctly assigned chest leads will be assessed (e.g. V4 is expected to be assigned to bV4)
Heart rhythm | 1 hour
  ECGs will be assessed for rhythm (eg. sinus rihythm, atrial fibrillation) by two board certified cardiologists
Ventricular depolarisation abnormalities | 1 hour
  ECGs will be assessed for ventricular depolarisation abnormalities (eg. bandle branch blocks) by two board certified cardiologists
Ventricular repolarisation abnormalities | 1 hour
  ECGs will be assessed for ventricular repolarisation abnormalities (eg. ST elevation) by two board certified cardiologists

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Universitiy Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No